CLINICAL TRIAL: NCT06323824
Title: Office-based Methadone Versus Buprenorphine to Address Retention in Medication for Opioid Use Disorder Treatment - A Pragmatic Hybrid Effectiveness/Implementation Trial
Brief Title: Office-based Methadone Versus Buprenorphine to Address Retention in Medication for Opioid Use Disorder Treatment.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry); University of California, San Francisco (Other); Boston Medical Center (BMC) (Unknown); Hennepin Healthcare Research Institute (Other); Alameda Health System (Other); Marshall Health (Unknown); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000033271; CTN-0131 (Other: Clinical Trials Network); 5UG1DA015831-21 (NIH)
Record Dates: First submitted 2023-03-13; First posted 2024-03-21 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder; Methadone; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone; Buprenorphine

STUDY DESIGN:
Intervention Model Description: The comparative effectiveness of two strategies to address retention in medication for opioid use disorder (MOUD) treatment will be tested over a 168-day period. Behavioral treatments offered to patients are designed to be similar across the two medication conditions.
  Office-based methadone where the clinician prescribes methadone and oral methadone is administered and/or dispensed at a pharmacy. Providers and Randomized Control Trial (RCT) participants will have flexibility to use behavioral and pharmacological services as clinically indicated.
  Office-based buprenorphine (BUP) where the clinician prescribes BUP formulations that are dispensed at a pharmacy or administered in the office (e.g., extended-release formulations). Providers and RCT participants will have flexibility to use behavioral and pharmacological services as clinically indicated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Office-based methadone (Experimental): Under special Drug Enforcement Administration (DEA) exception, Clinician prescribes methadone and oral methadone is administered and/or dispensed at a pharmacy which also has an exception to do so. All randomized controlled trial (RCT) participants are offered additional behavioral treatments (e.g., individual, group, telehealth, phone-based).
  Interventions: Drug: Methadone
- Office-based buprenorphine (BUP) (Active Comparator): Clinician prescribes BUP formulations that are dispensed at a pharmacy or administered in the office (e.g., extended-release formulations). All RCT participants are offered additional behavioral treatments (e.g., individual, group, telehealth, phone-based).
  Interventions: Drug: Buprenorphine (BUP)

INTERVENTIONS:
Drug: Methadone — Drug: Methadone
  Possible formulations:
  10 and 50 mg tablets
  Arms: Office-based methadone
Drug: Buprenorphine (BUP) — Drug: Buprenorphine (BUP)
  Possible formulations:
  A. Buprenorphine 225 mcg to 24 mg 225 mcg to 32 mg per day
  B. Buprenorphine (Extended release) 300 mg q 28 days (Sublocade) 100 mg q 28 days (Sublocade) 8 mg q 7 days (Brixadi) 16 mg q 7 days (Brixadi) 24 mg q 7 days (Brixadi) 32 mg q 7 days (Brixadi) 64 mg q 7 28 days (Brixadi) 96 mg q 7 28 days (Brixadi) 128 mg q 7 28 days (Brixadi)
  Arms: Office-based buprenorphine (BUP)

SUMMARY:
The purpose of this clinical trial is to compare the effectiveness of office-based methadone with pharmacy administration and/or dispensing to office-based buprenorphine for the treatment of opioid use disorder. This study will also examine factors influencing the implementation of office-based methadone.

DETAILED DESCRIPTION:
This study is a randomized, pragmatic hybrid type 1 effectiveness/implementation multisite (approximately 6 sites) trial to determine whether office-based methadone with pharmacy administration and/or dispensing or buprenorphine (BUP) results in greater treatment retention in approximately 600 patients with opioid use disorder (OUD). This trial will also identify implementation barriers, facilitators and acceptability at the patient, provider and health-systems level for office-based methadone with pharmacy administration and/or dispensing.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older;
* Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for OUD;
* Are initiating a new MOUD treatment episode

Exclusion Criteria

* Have been prescribed (and ingested) or been administered more than 72 hours of MOUD in the 7 days prior to randomization as a "bridge" to the new OUD treatment episode. Such MOUD may include prescribed (and ingested) or administered medically managed withdrawal (aka detoxification).
* Known contraindication to methadone or BUP
* Unwilling to pursue or continue pre-natal care or pregnancy counseling if determined pregnant by urine human chorionic gonadotropin (hCG) testing at the screening assessment
* Be actively suicidal or severely cognitively impaired (e.g., dementia, untreated psychosis) precluding informed consent as determined by site clinician
* Current severe comorbid substance use disorder requiring residential or inpatient treatment services as determined by site clinician
* Be unable to provide locator information including one or more contacts in addition to themselves
* Be unwilling to follow study procedures (e.g., unwilling to receive treatment from site clinician, use the study pharmacy, unwilling to be randomized to BUP or methadone, or will be unavailable for the follow-up assessments) including allowing the researchers to access their record in the EMR and state's prescription drug monitoring program
* Have previously enrolled in CTN-0131
* Currently enrolled in another research study which will conflict with study procedures
* Are currently in jail, prison or other overnight facility as required by a court of law or have pending legal action that could prevent participation in study activities
* Unable to conduct research assessments in English as determined by Site PI or their designee.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of days of continuous treatment with study site clinician-prescribed methadone or buprenorphine, as randomized, during the 168 days post-randomization among RCT participants. | up to Day 168
  MOUD dispensed to the participant including medication, duration of prescription and daily dose prescribed data will be extracted from the state prescription drug monitoring program (PDMP) and the electronic medical record (EMR).

SECONDARY OUTCOMES:
Number of self-reported days in any FDA-approved formulation of MOUD treatment (e.g., buprenorphine, methadone or naltrexone) during the 168 days post-randomization. | up to Day 168
  The MOUD Calendar Based Recall (Self-Report) form is used to collect self-reported prescribed medications for OUD.
Number of self-reported days in formal OUD treatment, according to American Society of Addiction Medicine (ASAM) levels of care 1-4, during the 168 days post-randomization. | up to Day 168
  This information will be obtained from one or more of the following:
  Health Services Utilization instrument, a brief structured interview regarding health care utilization (inpatient and outpatient) collecting information on the type and amount of services received, Timeline Followback Medications, MOUD Calendar Based Recall, and Treatment Dates instruments.
Number of days prescribed any FDA-approved MOUD formulation during the 168 days post-randomization. | up to Day 168
  MOUD dispensed to the participant including medication, duration of prescription and daily dose prescribed data will be extracted from the state prescription drug monitoring program (PDMP) and the electronic medical record (EMR).
Number of days of self-reported non-prescribed opioid use per month. | up to Day 168
  The Opioid Use Calendar Based Recall instrument is used to collect self-reported non-prescribed opioid use.
Number of days of self-reported non-prescribed stimulant use per month. | up to Day 168
  The Timeline Followback instrument collects self-reported drug and alcohol use.
Number of days of self-reported non-prescribed benzodiazepine use per month. | up to Day 168
  The Timeline Followback instrument collects self-reported drug and alcohol use.
Urine toxicology | up to Day 168
  Number of monthly urines negative for non-prescribed opioids during the 168 days post-randomization. Non-prescribed opioids will be determined using the Opioid Use Calendar Based Recall self-report.
Participant satisfaction with MOUD | up to Day 168
  Proportion of RCT participants who report at the assessment scheduled to be collected on day 28 that the medication they received was at least "Somewhat helpful" on the Satisfaction with MOUD Provider Scale instrument.
Total number of self-reported overdose events per total number of participant days at risk. | up to Day 168
  The Overdose Calendar Recall instrument collects overdose events.
Total number of self-reported injection drug use related events per total number of participant days at risk. | Up to Day 168
  Assessment of Infectious or Other Complications of Injection Drug Use assess for self-report of skin or soft-tissue infections, osteoarticular infections (septic arthritis, osteomyelitis, epidural abscess), endovascular infections including endocarditis, or new injection-related viral infections.
Pain measured using PEG-3: "Pain average," "interference with Enjoyment of life," and "interference with General activity." | Up to Day 168
  Mean scores on the PEG-3 screening instrument over time. Total score range is 0-10; the highest being the worse pain.
Number of self-reported days with acute care utilization (ED or hospitalization) events during the 168 days post-randomization per month. | Up to Day 168
  The Health Services Utilization instrument is a brief, structured interview regarding health care utilization (inpatient and outpatient) collecting information on the type and amount of services received. This includes ED visits, hospitalizations, primary medical care visits (excluding those for BUP treatment) and self-help sources of support (e.g., NA). Also assessed are receipt of formal and informal addiction and mental health treatment services RCT participants might have received outside the study interventions.

CONTACTS AND LOCATIONS:
Overall Officials: David Fiellin, MD, Principal Investigator — Yale University
Locations (6):
- United States (6):
  - Highland Hospital Bridge Clinic at Alameda Health System, Oakland, California
  - Outpatient Buprenorphine Induction Clinic, University of California, San Francisco, San Francisco, California
  - Rapid Start Clinic, Kaiser Permanente Colorado, Denver, Colorado
  - Officed Based Addiction Treatment Program, Boston Medical Center, Boston, Massachusetts
  - Hennepin Healthcare Addiction Medicine, Minneapolis, Minnesota
  - Marshall University Division of Addiction Sciences P.R.O.A.C.T, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
The National Institute on Drug Abuse (NIDA) Data Share web site is an electronic environment that allows data from completed clinical trials to be distributed to investigators and the public in order to promote new research, encourage further analyses, and disseminate information to the community. Secondary analyses produced from data sharing multiply the scientific contribution of the original research. NIH expects and supports the timely release and sharing of final research data from NIH-supported studies for use by other researchers to expedite the translation of research results into knowledge, products and procedures to improve human health.
Supporting Information: Study Protocol, SAP
Time Frame: Data sets will be available after (1) the primary paper has been accepted for publication, or (2) the data is locked for more than 18 months, whichever comes first.
Access Criteria: Public
URL: https://datashare.nida.nih.gov/